CLINICAL TRIAL: NCT04053660
Title: Effect Of Non-Surgical Periodontal Treatment On Endogenous Anti-Inflammatory Lipid Mediators In Patients With Chronic Periodontitis
Brief Title: Effect Of Non-Surgical Periodontal Treatment On Lipoxin a4 Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Ceren Gökmenoğlu, Principal invesitgator, Ordu University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Ordu dental faculty
Record Dates: First submitted 2019-08-02; First posted 2019-08-12 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Periodontitis
Keywords: Gingival Crevicular Fluid; Lipid Mediator; Periodontal Treatment
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Periodontally healthy group
- Chronic Periodontitis (Experimental): Patients with chronic periodontitis
  Interventions: Procedure: Non-surgical periodontal treatment

INTERVENTIONS:
Procedure: Non-surgical periodontal treatment — Mechanical non-surgical treatment were performed
  Arms: Chronic Periodontitis

SUMMARY:
The aim of this study was to evaluate the levels of lipoxin A4 (LXA4), prostaglandin E2 (PGE2) and leukotriene B4 (LTB4) in gingival crevicular fluid (GCF) and saliva in individuals with periodontal healthy and chronic periodontitis. In addition, the investigators evaluated the levels of these mediators after non-surgical periodontal treatment in patients with chronic periodontitis. A total of 20 subjects, 10 patients with chronic periodontitis (CP) and 10 periodontally healthy individuals were included in the study. Clinical parameters including plaque index (PI), gingival index (GI), probing depth (PD) and clinical attachment levels (CAL) were recorded. GCF and saliva samples were obtained at the beginning of the study from all individuals. GCF and saliva samples were re-collected from patients with CP at 1 month after non surgical periodontal therapy.

ELIGIBILITY:
Inclusion Criteria:

* Have at least 20 natural teeth, excluding third molars.
* Chronic periodontitis patients had at least two non-adjacent sites per quadrant with probing depth (PD) ≥ 5 mm and clinical attachment level (CAL) ≥ 5 mm with gingival inflammation, and alveolar bone loss affecting >30% of the teeth, as detected on clinical and radiographical examinations.
* Periodontally healthy control group had no sign of gingival inflammation, no PD > 3mm and no evidence of attachment or bone loss.

Exclusion Criteria:

* History of systemic disease.
* Regular use of any drugs which can effect the immune system or inflammatory response in the 6 months preceding the start of the study.
* Periodontal treatment during last 6 months that could affect periodontal status.
* Smoking.
* History of radiotherapy or chemotherapy.
* Ongoing orthodontic treatment.
* Aggressive periodontitis.
* Current pregnancy, lactation or menopause.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Lipoxin A4 levels | 1st month
  change of gingival crevicular fluid and salivary Lipoxin A4 levels from baseline at 1st month

SECONDARY OUTCOMES:
Prostaglandin E2 levels | 1st month
  change of gingival crevicular fluid and salivary Prostaglandin E2 levels from baseline at 1st month
Leukotriene B4 | 1st month
  change of gingival crevicular fluid and salivary Leukotriene B4 levels from baseline at 1st month

CONTACTS AND LOCATIONS:
Overall Officials: Ceren Gokmenoglu, Principal Investigator — Ordu University Faculty of Dentistry
Locations (1):
- Ordu University, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No